Local dishes versus 'ready-to-use therapeutic foods' in the management of severe acute malnutrition during the rehabilitation phase: a randomized, single-blind study at the regional hospital annex of Mokolo (Cameroon)

ID: 062/24L/MSP/DRSP-EN/HRA-MOK

NCT ID (In process)

| INFORMED CONSENT FORM |
|---|
| I, the undersigned |
| declare to accept, freely, and in an informed manner to participate as a subject in the stud |
| entitled: EFFECTIVENESS OF ENHANCED AWARENESS ON THE USE OF LOCA |
| DISHES AMONG SEVERELY ACUTE MALNOURISHED INDIVIDUALS I |
| REHABILITATION AT THE REGIONAL HOSPITAL ANNEX OF MOKOLO. |
| Under the direction of: Prof. SAP SUZANNE, Dr. KAMO HELENE, and Dr. FADIMATO |
| ALTINE |
| Promoter: University of Garoua (Faculty of Medicine and Biomedical Sciences of Garoua) |
| Principal Investigator: SEPTCHE DAVY GILLES, 7th-year student |
| Commitment of the principal investigator: as the principal investigator, he commits |
| conducting this research according to ethical and deontological provisions, to protect the |
| physical, psychological, and social integrity of individuals, and to ensure the confidentiality |
| the information collected. He also commits to providing participants with all the support |
| mitigate any negative effects that may arise from participation in this research. |
| Participant's freedom: consent to continue the research can be withdrawn at any time witho |
| giving a reason and without incurring any liability or consequence. Responses to questions a |
| optional, and failure to respond will have no consequences for the subject. |
| Participant information: the participant has the opportunity to obtain additional information |
| regarding this study from the principal investigator, within the limits of the constraints of the |
| research plan. |
| Confidentiality of information: all information concerning participants will be kept anonymou |
| and confidential. The computer processing is not nominative; thus, it does not fall under the |

data protection law (the right of access and rectification is not applicable). The transmission of information concerning the participant for expertise or scientific publication will also be anonymous.

| Deontology | and et | hics: tl | ne prom | oter and | d the | investigator | commit | to | absolutely | preserving |
|---|---|---|---|---|---|---|---|---|---|---|
| confidentiality and professional secrecy for all information concerning the participant. | | | | | | | | | | |

| Done at | on | <br> | ••• | ••• | • • • | <br> |
|-------------|----|------|-----|-----|-------|------|
| In 2 copies | | | | | | |

The participant.

The principal investigator.